CLINICAL TRIAL: NCT00334737
Title: A Randomized, Masked, Placebo Controlled Study to Assess the Safety and Efficacy of Darbepoetin Alfa Administered to Preterm Infants
Brief Title: Darbepoetin Administration to Preterm Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Thrasher Research Fund (Other); University of Colorado, Denver (Other); Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-139
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Infant, Newborn
Keywords: erythropoietin; darbepoetin; transfusions; neonates; outcomes; neurodevelopment
MeSH Terms: interventions — Darbepoetin alfa; Epoetin Alfa; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Darbepoetin alfa injection (Experimental): Darbepoetin alfa 10 mics/kg/week subcutaneous injection x 10 weeks or until 35 completed weeks Drug: Darbepoetin alfa Other names: Aranesp Darbe SC injection
  Interventions: Drug: Darbepoetin Alfa Injection
- erythropoietin alfa injection (Active Comparator): Epo 400 units/kg three times a week SC x 10 weeks or until 35 completed weeks Drug: erythropoietin other names: epogen Epo SC injection
  Interventions: Drug: erythropoietin alfa injection
- placebo/control (Placebo Comparator): Sham injection
  Interventions: Drug: sham injection

INTERVENTIONS:
Drug: Darbepoetin Alfa Injection — darbepoetin alfa injection 10 mics/kg once a week SC for 10 weeks or until 35 completed weeks
  Other Names: aranesp; Darbe
  Arms: Darbepoetin alfa injection
Drug: erythropoietin alfa injection — Epo 400 units/kg 3 x weekly SC for 10 weeks or until 35 completed weeks gestation
  Other Names: procrit, epoetin alfa
  Arms: erythropoietin alfa injection
Drug: sham injection — sham injection other names: not applicable
  Other Names: placebo
  Arms: placebo/control

SUMMARY:
Infants born prematurely do not increase production of the primary red cell growth factor, erythropoietin (Epo), and often develop an anemia called the "anemia of prematurity." The anemia of prematurity is the most common anemia seen in neonates, and is due to a failure of Epo production. Human recombinant Epo (rHuEpo), given three to five times a week, is successful in treating the anemia of prematurity. A slightly modified, long-acting version of rHuEpo, called darbepoetin alfa (darbepoetin), is now available and has proven effective in increasing hematocrit (red blood cell levels) in adults. In addition to its red cell stimulating properties, recent evidence has shown that rHuEpo is protective in the developing or injured brain. We have designed a randomized, masked, placebo-controlled study to determine the safety and short and long term efficacy of darbepoetin. At this time, darbepoetin has been studied primarily in adults and pediatric patients, but there is evidence from pilot studies that darbepoetin would be useful in the neonatal setting as well. It also may well improve neurodevelopmental outcomes in preterm neonates. We hypothesize that: 1. The administration of darbepoetin to preterm infants 500 to 1,250 grams birth weight will result in increased reticulocyte counts and decreased transfusions compared to placebo; and 2. The administration of darbepoetin will be associated with an increased mental developmental index at 18-22 months compared to placebo.

DETAILED DESCRIPTION:
A novel erythropoiesis stimulating protein, Darbepoetin alfa (Darbepoetin) has been developed by Amgen Inc. and has been shown to be effective in increasing hematocrit using once weekly or once every other week dosing in adults with anemia due to end stage renal disease or cancer. However, it is presently being evaluated for use in children with hyporegenerative anemias, and has not yet been evaluated for use in infants with anemia of prematurity. Preterm infants respond to human recombinant erythropoietin (Epo) by increasing reticulocytes, yet the multiple subcutaneous doses diminish its routine use in the NICU. With the possibility of once a week or once every other week dosing, the use of Darbepoetin in this population appears promising. While it is likely that the use of red cell growth factors such as rHuEpo or darbepoetin will not eliminate the need for all erythrocyte transfusions in all infants, it is reasonable to postulate that the use of darbepoetin will eliminate the need for transfusion in some preterm infants, and reduce the need in others. European studies evaluating rHuEpo in preterm infants have successfully decreased donor exposure to 1 per patient. Our goal is to achieve similar success, which we define as a donor exposure of ≤1 donor per infant in clinical practice. This can be achieved through the use of red cell growth factors, judicious use of blood work for monitoring, and stringent transfusion guidelines. By decreasing total transfusions to <4 per infant, we can achieve this goal of ≤1 donor exposure per infant.

There will remain a population of extremely small, extremely ill infants in whom phlebotomy losses exceed the capacity to increase red cell mass through the use of Epo. Some investigators believe a combination of single donor erythrocyte transfusions and recombinant erythropoietin can serve to maintain an adequate circulating erythrocyte volume. A reasonable algorithm can be developed to assist in these determinations only through continued research. Continued critical evaluation of transfusion criteria, outcomes, new technologies limiting phlebotomy loss, and novel biologic and pharmacologic treatments can only serve to improve the care of ELBW infants who are highest risk for repeated transfusions. Our research aim is to study the safety and efficacy of darbepoetin in preterm infants in order to improve the outcomes of preterm infants by significantly decreasing the number of transfusions. Moreover, improving neurodevelopmental outcomes for preterm infants continues to be a goal for neonatal care providers that might begin to be approached through darbepoetin therapy. This study differs from previous erythropoietin studies in the following ways:

1. Darbepoetin will be compared to placebo and to rHuEpo, allowing two thirds of the patients to receive some form of red cell growth factor, and allowing SC dosing to occur once a week in the darbepoetin recipients compared with the usual three times a week SC dosing in the rHuEpo recipients (those in the placebo group will not receive sham injections)
2. Dosing will begin 1-2 days earlier on average than in any previously published study
3. Transfusion guidelines are the most rigorous applied to date, and will be used at sites that are all at altitudes > 4,000 feet
4. A target Epo concentration of >500 mU/mL in the treatment group is proposed in order to evaluate neurodevelopmental differences between groups, and the study is powered to determine a difference between treatment groups and placebo

ELIGIBILITY:
Inclusion Criteria:

* 500-1250 grams birth weight
* less than or equal to 32 weeks gestation
* less than 2 days of age

Exclusion Criteria:

* severe hemorrhagic disease
* severe hemolytic disease
* DIC
* seizures
* hypertension
* thromboses
* receiving erythropoietin

Ages: 1 Hour to 49 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2006-06; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin K Ohls, MD, Principal Investigator — University of New Mexico; Robert D Christensen, MD, Principal Investigator — McKay-Dee Hospital, Ogden, Utah; Susan Wiedmeier, MD, Principal Investigator — LDS Hospital, Salt Lake City, Utah; Adam Rosenberg, MD, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - McKay-Dee Hospital, Ogden, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Will enter in DASH if appropriate

REFERENCES:
- [Background] Warwood TL, Ohls RK, Wiedmeier SE, Lambert DK, Jones C, Scoffield SH, Neeraj G, Veng-Pedersen P, Christensen RD. Single-dose darbepoetin administration to anemic preterm neonates. J Perinatol. 2005 Nov;25(11):725-30. doi: 10.1038/sj.jp.7211387. PMID 16151471
- [Background] Ohls RK, Dai A. Long-acting erythropoietin: clinical studies and potential uses in neonates. Clin Perinatol. 2004 Mar;31(1):77-89. doi: 10.1016/j.clp.2004.03.006. PMID 15183658
- [Background] Warwood TL, Ohls RK, Lambert DK, Jones C, Scoffield SH, Gupta N, Veng-Pedersen P, Christensen RD. Intravenous administration of darbepoetin to NICU patients. J Perinatol. 2006 May;26(5):296-300. doi: 10.1038/sj.jp.7211498. PMID 16554846
- [Background] Ohls RK, Ehrenkranz RA, Das A, Dusick AM, Yolton K, Romano E, Delaney-Black V, Papile LA, Simon NP, Steichen JJ, Lee KG; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcome and growth at 18 to 22 months' corrected age in extremely low birth weight infants treated with early erythropoietin and iron. Pediatrics. 2004 Nov;114(5):1287-91. doi: 10.1542/peds.2003-1129-L. PMID 15520109
- [Derived] Lowe JR, Rieger RE, Moss NC, Yeo RA, Winter S, Patel S, Phillips J, Campbell R, Baker S, Gonzales S, Ohls RK. Impact of Erythropoiesis-Stimulating Agents on Behavioral Measures in Children Born Preterm. J Pediatr. 2017 May;184:75-80.e1. doi: 10.1016/j.jpeds.2017.01.020. Epub 2017 Feb 6. PMID 28185625
- [Derived] Ohls RK, Cannon DC, Phillips J, Caprihan A, Patel S, Winter S, Steffen M, Yeo RA, Campbell R, Wiedmeier S, Baker S, Gonzales S, Lowe J. Preschool Assessment of Preterm Infants Treated With Darbepoetin and Erythropoietin. Pediatrics. 2016 Mar;137(3):e20153859. doi: 10.1542/peds.2015-3859. Epub 2016 Feb 15. PMID 26908704

RESULTS

PARTICIPANT FLOW:
Groups:
- Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w: Darbepoetin 10 mics/kg/week x 10 weeks or until 35 completed weeks
  darbepoetin alfa: darbepoetin 10 mics/kg once a week SC for 10 weeks or until 35 completed weeks
- Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35: Epo 400 units/kg three times a week SC x 10 weeks or until 35 completed weeks
  erythropoietin: Epo 400 units/kg 3 x weekly SC for 10 weeks or until 35 completed weeks gestation
- Placebo/Control: Sham injection
  sham injection: sham injection
Period: Hospital Phase
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Started | 34 | 34 | 34
Completed | 32 | 32 | 30
Not Completed | 2 | 2 | 4
Not completed — Death | 1 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Did not receive study drug | 1 | 0 | 0
Period: Follow up Phase
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Started | 32 | 32 | 30
Completed | 27 | 29 | 24
Not Completed | 5 | 3 | 6
Not completed — Lost to Follow-up | 5 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control | Total
Number analyzed (Participants) | 27 | 29 | 24 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 20 [20 to 21] | 21 [20 to 22] | 20 [19.5 to 21] | 21 [20 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 9 | 36
  Male | 10 | 19 | 15 | 44
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 24 | 80
gestation [Median (Inter-Quartile Range); unit: weeks] | 28.3 [26.5 to 29.5] | 27.7 [26.2 to 29.1] | 28.1 [27.1 to 28.8] | 28 [26.5 to 28.9]
birthweight [Median (Inter-Quartile Range); unit: grams] | 980 [801 to 1090] | 930 [778 to 1158] | 1005 [810 to 1133] | 975 [800 to 1135]

OUTCOME MEASURES:

1. Primary Outcome: Number of Transfusions During Hospitalization
Time Frame: From birth to 36 weeks gestational age
Measure: Mean (Standard Deviation); unit: number of transfusions
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 33 | 33 | 33
number of transfusions | 1.2 (2.4) | 1.2 (1.6) | 2.4 (2.9)

2. Primary Outcome: Composite Cognitive Score at 18-22 Months Corrected Age
Description: Bayley Scale of Infant Development Composite Cognitive Score. The total composite score is reported, ranging from the lowest score of 55 to the highest score of 145. Lower values specify worse outcome.
Time Frame: 18-22 months
Measure: Mean (Standard Deviation); unit: BSID III compositie cognitive score
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 27 | 29 | 24
BSID III compositie cognitive score | 96.2 (7.2) | 97.9 (14.3) | 88.7 (13.5)

3. Secondary Outcome: Hematocrit
Time Frame: From birth to 36 weeks gestational age
Measure: Mean (Standard Deviation); unit: L/L
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 32 | 32 | 30
L/L | 0.35 (0.09) | 0.36 (0.08) | 0.29 (0.09)

4. Secondary Outcome: Reticulocyte Count
Description: absolute retic count measured at the end of study
Time Frame: at day 60 of study
Measure: Mean (Standard Error); unit: 1000 cells per microliter
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 32 | 32 | 30
1000 cells per microliter | 295 (50) | 298 (47) | 130 (70)

5. Secondary Outcome: Volume of Transfusions
Time Frame: From birth to 36 weeks gestational age
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 32 | 32 | 30
mL/kg | 30 (58) | 23 (33) | 51 (65)

6. Secondary Outcome: Epo Concentrations
Time Frame: peak from birth to 36 weeks gestational age
Population: One hospital participating in the trial lost their samples. The number analyzed only includes those with samples.
Measure: Mean (Standard Deviation); unit: mU/mL
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 19 | 16 | 20
mU/mL | 1398.9 (882.7) | 515.4 (280.3) | 28.6 (51.1)

7. Secondary Outcome: Object Permanence Scores at 18-22 Months
Description: Scores are 0-3, with 3 being the best score.
Time Frame: 18-22 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 27 | 29 | 24
units on a scale | 2.8 (0.4) | 2.4 (0.9) | 2.2 (1.0)

8. Secondary Outcome: Overall Neurodevelopmental Impairment at 18-22 Months (Visual Impairment, Hearing Impariment, Cerebral Palsy, or Cognitive Score <85/<70 (NDI/Moderate NDI)
Time Frame: 18-22 months
Measure: Number; unit: participants
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 28 | 30 | 27
participants | 4 | 5 | 13

9. Secondary Outcome: Incidence of Retinopathy of Prematurity Stage 3 or Greater
Time Frame: From birth to 36 weeks gestational age
Measure: Number; unit: participants
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Number analyzed (Participants) | 32 | 32 | 30
participants | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: Initial hospitalization after preterm birth
Description: Adverse events collected during subject's initial hospitalization in the NICU
Arm/Group | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 | Placebo/Control
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/33 | 3/33
Other Adverse Events (participants affected / at risk) | 5/33 | 4/33 | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w (N=33) | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 (N=33) | Placebo/Control (N=33)
death (General disorders) | 1 (33) | 1 (33) | 3 (33) — mortality during initial hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Darbepoetin 10 Mics/kg/Week x 10 Weeks or Until 35 Completed w (N=33) | Epo 400 Units/kg Three Times a Week SC x 10 Weeks or Until 35 (N=33) | Placebo/Control (N=33)
ROP>stage 2 (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
IVH>grade 2 (Nervous system disorders) | 3 (3) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No